CLINICAL TRIAL: NCT04221776
Title: Implementing a New Method of Group Toilet Training in Daycare Centers: a Cluster Randomised Controlled Trial
Brief Title: Group Toilet Training of Healthy Children, in Daycare Centers (CRCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Tinne Van Aggelpoel, Pelvic floor physiotherapist, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B300201630079
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Toilet Training; Child, Preschool
Keywords: Method
MeSH Terms: interventions — Child Day Care Centers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive toilet training group (Experimental): Intervention group was subjected to an intensive TT group session lasting 2-hours during 2 consecutive days in daycare centers.
  Interventions: Other: Group toilet training in daycare
- Standard care toilet training group (Active Comparator): Children participating in control group did not receive the intensive training, but parents got a leaflet and were encouraged to start TT their child at home, in their own manner.
  Interventions: Other: Individual toilet training at home

INTERVENTIONS:
Other: Group toilet training in daycare — During the training, children wore underpants, were informed about potty training, were encouraged to drink often and were asked regularly if they felt the need to void. Tutors looked for elimination signals in the child and quickly responded by putting the child on the potty when he/she expressed the need to void or to defecate. Children were positively rewarded. Parents received a leaflet containing practical tips concerning TT and their child's successes of the past two days. They were asked to continue TT at home during the following weekend and longer if necessary. Daycare workers were asked to pay more attention on the TT during the following days and weeks to ensure the effect of the intervention.
  Arms: Intensive toilet training group
Other: Individual toilet training at home — Parents were encouraged to start TT their child, because they were considered as being ready to initiate TT. Children did not receive any intervention, but parents were asked to start TT in their own manner. Parents were allowed to search for information on methods of TT with their relatives, internet, books,...
  Arms: Standard care toilet training group

SUMMARY:
Evaluation of a new method of toilet training (TT), meaning TT in group in daycare centers, guided by a TT expert. Children are included based on signs of readiness for TT.

DETAILED DESCRIPTION:
A cluster randomized controlled trial (CRCT) was established in daycare centers. Clusters of participants (per daycare center) were randomly allocated to an Intervention group or a Control group.

Evolution of the TT process was monitored in the daycare center until the child was considered to be fully toilet trained (or 'clean') during the day (this means wearing undergarments, conscious of the need to void and initiating toilet behavior without reminder of the parents with a maximum of one leakage a day [9]).

Daycare workers evaluated the TT process of all participating children on a weekly basis. Parents were asked to fill in an online questionnaire when their child was completely toilet trained.

ELIGIBILITY:
Inclusion Criteria:

* knowledge of the Dutch language
* aged between 18 and 30 months
* not yet toilet trained during the day and night (diaper dependent)
* Parents of the children had to be motivated to participate in the study and willing to invest time and effort in continuing the TT at home
* Children met at least two of the following three signs of readiness: the child expresses a need to evacuate and shows awareness of the need to void or to have a bowel movement; the child insists on completing tasks without help and is proud of new skills; or the child can pull clothes up and down in a TT related context

Exclusion Criteria:

* Children with urological, neurological, organical or behavior problems

Ages: 18 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Duration of toilet training | 6 weeks
  Number of weeks needed for the child to become fully toilet trained

SECONDARY OUTCOMES:
Effectiveness of toilet training | 6 weeks
  Number of children that acquire cleanliness at 6 weeks time

CONTACTS AND LOCATIONS:
Overall Officials: Van Aggelpoel, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Aggelpoel T, De Wachter S, Neels H, Van Hal G, Roelant E, Vermandel A. Implementing a new method of group toilet training in daycare centres: a cluster randomised controlled trial. Eur J Pediatr. 2021 May;180(5):1393-1401. doi: 10.1007/s00431-020-03879-y. Epub 2020 Nov 23. PMID 33230718